CLINICAL TRIAL: NCT03920592
Title: Effect of Bullying Content Presented in Immersive 360º-video on Pupil's Cognitive and Psychophysiological Responses
Brief Title: Virtual Reality and Prevention of Bullying
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Narcis Cardoner, MD, PhD (Other)
Collaborators: Fundació Eurecat (Other); Recercaixa (Unknown); Escola Parc del Guinardó (Unknown); Fundació FC Barcelona (Unknown)
Responsible Party: Sponsor-Investigator, Narcis Cardoner, MD, PhD, Psychiatrist, Director Depression and Anxiety Program & OSAMCAT, Corporacion Parc Tauli
Organization: Corporacion Parc Tauli (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: CSMPT_NC_2019_1
Record Dates: First submitted 2019-04-09; First posted 2019-04-19 (Actual); Last update posted 2019-04-29 (Actual); Status verified 2019-04

CONDITIONS: Bullying of Child
Keywords: Virtual reality; Psychophysiology; Empathy

STUDY DESIGN:
Intervention Model Description: Each participant, depending on their sex, watch two minutes of each video content:
  1. Bullying content in virtual reality
  2. Bullying content in a regular 2D screen
  3. Pupils playing without bullying content in virtual reality
  4. Pupils playing without bullying content in a regular 2D screen
Masking Description: Participants are unaware of which condition is being tested
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Video watching (Experimental): All participants will watch 4 videos of potential everyday school situations, adapted for boys and girls.
  Videos contain different levels of bullying (presence/absence) and virtual reality (presence/absence).
  Every pupil will watch the 4 types of video content randomly.
  Interventions: Behavioral: Virtual Reality of Bullying

INTERVENTIONS:
Behavioral: Virtual Reality of Bullying — Immersive videos (360º) filmed by 12-14 year old pupils who, guided by professional actors, represented the subjective experience of bullying.
  Eight different potential situations designed depending on the sex of the pupil were filmed:
  Girls:
  1. Classmates steal her personal diary
  2. Classmates tear her clothing
  3. Classmates insult her and steal her belongings
  4. Classmates deliberately exclude her in class
  Boys:
  1. Classmates exclude him while playing with a ball
  2. Classmates bother him in the dining room
  3. Classmates insult and steal him in class
  4. Classmates insult him and steal his belongings

SUMMARY:
The lack of empathy towards victims of bullying is thought to play a main role in this extended and pernicious peer victimization behaviour. Thus, promoting empathy in school programs might be a promising approach for bullying prevention. Virtual reality (VR) allows creating an environment very similar to the real world and has proved to promote empathy.

Therefore, by employing VR, pupils may better understand and feel the experience of being bullied. As there is no evidence of the efficiency of VR in bullying prevention, the first step is to validate the content of the environments created.

In this line, the current study aims to investigate if 360º-videos produce a truthful experience of being bullied superior than the observed in traditional computer screens. The effect of all, 360º-videos and 2D computer screens will be assessed through objective (electrodermal activity -EDA- and heart rate -HR-) and subjective (self-administered tests) measures.

DETAILED DESCRIPTION:
Introduction and Rationale: Previous research suggests that working on the development of cognitive-emotional skills, and particularly on empathy toward victims of bullying, may be a central component for the success of school bullying prevention programs. On the other hand, virtual reality (VR) technology allows adopting the perspective of the world of others, and thus has been claimed to be a powerful tool for eliciting empathy in different domains (cf. Slater & Sánchez-Vives, 2016). Therefore, VR might play a role in bullying prevention programs, by helping pupils to understand how it feels to be bullied, as a way to increase empathy towards victims of bullying. However, currently empirical evidence of the effectiveness of VR in this context is lacking. A key step in the validation of this use of VR is to understand how the immersive presentation of bullying scenes shot from a first-person perspective is experienced by children, compared to the same scenes presented in less immersive displays. In particular, in order to demonstrate the potential of VR technology in this regard, it is necessary to examine the advantages that VR technology (and, more specifically in this case, immersive presentation of 360º-video) presents over more common devices (a computer screen).

Study goals and Hypotheses: The overall goal of this study is to examine whether 360º-videos representing situations of bullying from a first-person perspective produce a realistic experience of being bullied, and that the presentation of such contents in an immersive mode (using a VR headset) elicit a more realistic and arousing experience than the same contents in a less immersive format (a traditional computer screen).

This is the first step in a wider research project; in subsequent steps, the investigators will assess the effects of these type of videos on empathy towards victims of bullying and, eventually, on prevalence of bullying behaviour.

The central hypotheses to be tested will be:

Hypothesis 1 (H1): Contents representing situations of bullying from a first person perspective will elicit on participants realistic feelings of being bullied, compared to contents representing other high-school daily situations not involving (physical or verbal) violence.

Hypothesis 2 (H2): Immersive presentation (i.e. 360º-video contents watched in a VR headset) will elicit higher arousal and higher perceived realism of the scene than the same contents presented in a less immersive display (a computer screen).

In order to test these hypotheses, the investigators will collect measures of psychophysiological measures of arousal (electrodermal activity -EDA- and heart rate -HR-) and emotional regulation (heart rate variability -HRV-), self-reported emotional arousal and valence, as well as three self-reported measures of the realism of the experience of being bullied, including: (1) participant's perception on to which degree the represented situation can be considered bullying, (2) participant's feelings of actually being in the represented scene ("presence"), and (3) participant's feeling of actually being bullied while watching the content.

The investigators expect that, compared to watching videos representing other high-school daily situations not involving (physical or verbal) violence, watching videos representing situations of bullying, participants' EDA, HR, HRV, and self-reported arousal will be higher (H1a, H1b, H1c, and H1d, respectively), self-reported valence will be more negative (H1e), scores of feelings of being bullying and actually being in the scene will be higher (H1f and H1g, respectively), and the perception of the scene as bullying will also be enhanced (H1h).

It is also expected that, compared to the videos presented in a screen, while watching the videos in a VR headset participants' EDA, HR, HRV, and self-reported arousal will be higher (H2a, H2b, H2c, and H2d, respectively), self-reported valence will be more negative (H2e), scores of feelings of being bullying and actually being in the scene will be higher (H2f and H2g, respectively), and the perception of the scene as bullying will also be enhanced (H2h).

In addition, it will be explored whether the experienced arousal and perception of realism is associated with personality traits, such as being uncaring, unemotional, and callousness. The investigators believe that pupils with higher scores on the mentioned traits will experience less arousal (subjective and psychophysiological) when watching the videos with bullying content.

Experimental design: The study adopts a within-subject design in which each participant will watch four videos, containing the four possible combinations of two independent variables: Level of immersion (VR headset / computer screen) and Type of content (Bullying / no-bullying content).

The materials to be used in the experiment will be eight videos representing different scenes from the perspective of a girl (to be watched by female participants) and four videos representing different scenes from the perspective of a boy (to be watched by male participants). Among each group of eight videos, there are four pairs. The two videos of each pair involve the same location, point-of-view, and actors, but in one of them there is a bullying situation and in the other there is a daily situation not involving any form of violence (e.g. children chatting about the last weekend).

Each participant will watch four scenes, two containing bullying scenes and the other containing daily non-violent scenes. Also, two of them will be presented in a VR headset while the rest be presented in a computer screen. The level of immersion and type of content in which each scene is presented will vary among participants following a Latin-square design, in a way such for the whole sample of participants, all the scenes will be presented across the two levels of immersion and the two types of content. The order of the presentation of the four conditions will be randomised for each participant.

ELIGIBILITY:
Inclusion Criteria:

* All pupils assisting 5th and 6th grade of primary school (Spain education system) of the "Escola Parc del Guinardó" school
* Pupils whos parents have read, understand and approved the informed consent of the study.

Exclusion Criteria:

* Pupils whose parents have not approved their inclusion in the study.

Ages: 9 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 34 (Actual)
Dates: Start 2019-04-10 (Actual); Primary Completion 2019-04-12 (Actual); Study Completion 2019-04-12 (Actual)

PRIMARY OUTCOMES:
Self-assessment manikin (SAM) | Baseline
  Arousal and valence (5-point graphic scale)
Heart rate (HR) and heart rate variability (HRV) | Baseline
  An electrocardiogram will be recorded as an indirect indicator of the physiological arousal.
Electrodermal activity (EDA) | Baseline
  The skin conductance will be registered as an indirect indicator of the physiological arousal. Tonic and phasic measures will be registered.

SECONDARY OUTCOMES:
The Inventory of Callous-Unemotional Traits (ICU) in Children | Baseline
  The self-report version of the ICU assesses uncaring, unemotional, and callousness traits.
  Te scale has 24-items, ranked on a 4-point Likert scale, from 0 (not at all true) to 3 (definitely true). Possible scores ranges from 0-72, where higher scores indicate greater presence of the construct.
Empathy toward victim | Baseline
  7-item scale to assess empathy towards bullying. Higher scores indicate greater presence of the construct.
Ad-hoc items regarding bullying | Baseline
  Two ad-hoc items on how much the video presents a situation of "bullying", and to which extent the participant feel "been bullied" while watching the video. 5-point Likert scale in which 0 means "none" and 5 "absolutely". The items were:
  1. I think the video represents a situation of harassment
  2. I have really felt harassed while looking at the video
Ad-hoc item on "presence" | Baseline
  Feeling of being involved in the virtual environment. 5-point Likert scale in which 0 means "none" and 5 "absolutely". The item was:
  3. I felt that I was "there" in the video scene

CONTACTS AND LOCATIONS:
Overall Officials: Narcís Cardoner, MD, PhD, Principal Investigator — Corporacion Parc Tauli; Miguel Barreda, PhD, Principal Investigator — Eurecat, Centre Tecnològic de Catalunya
Locations (1):
- Corporació Sanitària Parc Taulí, Sabadell, Spain

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fanti, K. A., & Kimonis, E. R. (2012). Bullying and Victimization: The Role of Conduct Problems and Psychopathic Traits. Journal of Research on Adolescence, 22(4), 617-631.
- [Background] Moore AA, Carney D, Moroney E, Machlin L, Towbin KE, Brotman MA, Pine DS, Leibenluft E, Roberson-Nay R, Hettema JM. The Inventory of Callous-Unemotional Traits (ICU) in Children: Reliability and Heritability. Behav Genet. 2017 Mar;47(2):141-151. doi: 10.1007/s10519-016-9831-1. Epub 2016 Dec 1. PMID 27909830
- [Background] Nickerson AB, Mele D, Princiotta D. Attachment and empathy as predictors of roles as defenders or outsiders in bullying interactions. J Sch Psychol. 2008 Dec;46(6):687-703. doi: 10.1016/j.jsp.2008.06.002. Epub 2008 Jul 15. PMID 19083379
- [Background] Munoz LC, Qualter P, Padgett G. Empathy and bullying: exploring the influence of callous-unemotional traits. Child Psychiatry Hum Dev. 2011 Apr;42(2):183-96. doi: 10.1007/s10578-010-0206-1. PMID 20886285